CLINICAL TRIAL: NCT04144478
Title: Web-Based Epilepsy Education Program for Adolescents and Parents: A Randomized Controlled Trial
Brief Title: Web-Based Epilepsy Education Program for Adolescents and Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Şerife TUTAR GÜVEN, Pediatric Nursing, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Suleyman Demirel University
Record Dates: First submitted 2019-10-17; First posted 2019-10-30 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; Web based education; Pediatric Nursing; Parent; Adolescence
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Web based education intervention
  Interventions: Other: Web based education
- No intervention (No Intervention): Normal polyclinics application

INTERVENTIONS:
Other: Web based education — Web based education
  Arms: experimental

SUMMARY:
This study aims to develop a web-based epilepsy education program for adolescents with epilepsy and their parents and to evaluate the efficacy of eb-based epilepsy education program on health management.eb-based epilepsy education program has been proved to be a useful and reliable educational website for the development of knowledge, attitude, self-efficacy and e-health literacy of adolescents with epilepsy and their parents.

DETAILED DESCRIPTION:
This study aims to develop a web-based epilepsy education program for adolescents with epilepsy and their parents and to evaluate the efficacy of web-based epilepsy education program on health management.

This randomized controlled study was conducted with 69 adolescents with epilepsy aged between 9-18 and their parents (n=71) who were accepted to Pediatric Neurology Policlinic of Antalya Training and Research Hospital of Health Science University between November 2017 and April 2018. The study sample was divided into two groups as study (35 adolescents, 37 parents) and control (34 adolescents, 34 parents) groups using simple randomization method. The web-based epilepsy training program which was developed during the preparation stage of the study was evaluated by 13 experts using the Quality of Criteria for Consumer Health Information measurement instrument. The data collection materials (Seizure Self efficacy scale, E-Health literacy scale, Child Attitude Toward Illness Scale, Website Analysis and MeasureMent Inventory Scale) were administered by the researcher to the adolescents and parents in both groups before applying eb-based epilepsy education program. Following the administration of eb-based epilepsy education program to the initiative group, all participants were observed for three months. The data collection materials were reapplied to all the participants at the end of the third month. In addition, the adolescents and their parents in the study group were applied Website Analysis and Measurement Inventory measurement tool for the evaluation of usability of the site.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents without mental disability,
* Followed-up for at least six months with epilepsy diagnosis,
* No chronic disease other than epilepsy,
* No photosensitive epilepsy diagnosis,
* Internet access and use, and parents of these adolescents with internet access and use - were included in the study.

Exclusion Criteria:

* Adolescents and parents who do not use the Internet

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Epilepsy Knowledge Test | 12 week
  Epilepsy Knowledge test had applied pre-test and post-test. It consists of true (1), false (0) and I do not know (0) options. The minimum score to be taken from the scale is 0 and the maximum score is 25. The minimum score to be taken from the scale is 0 and the maximum score is 25. The increase in the total score indicates that the level of knowledge has increased.
Seizure Self Efficacy Scale | 12 week
  Seizure Self Efficacy Scale had applied pre-test and post-test. The scale is a 5-point likert with 15 items. It has been interpreterd that the higher the total score, the higher is the self-efficacy level of the individual. The minimum score to be taken from the scale is 15 and the maximum score is 75.
Child Attitude Toward Ilness Scale | 12 week
  Child Attitude Toward Ilness Scale had applied pre-test and post-test. The scale was a 5-point Likert type with 15 items. The minimum score to be taken from the scale is 15 and the maximum score is 75. 25. The minimum score to be taken from the scale is 0 and the maximum score is 25. The increase in the total score indicates that the child has positive attitude own illness.
e-Health Literacy Scale | 12 week
  e-Health Literacy Scale had applied pre-test and post-test. The lowest score that can be obtained from the 5-point Likert scale is 8 and the highest score is 40. A high score from the scale indicates a high level of e-health literacy.
Website Analysis and MeasureMent Inventory | 12 week
  Website Analysis and MeasureMent Inventory had applied both website under preparation and post test for control group.There are 5 dimensions that measure concepts like Attractiveness, Controllability, Efficiency, Helpfulness and Learnability. The total usability score is the weighted combination of expressions from each of the five sub-dimensions. The higher the scores obtained from the scale, the higher is the usability of the website and the more useful it is. The score obtained from the Website Analysis and MeasureMent Inventory is calculated in percentiles. the fact that each sub-dimension is above 50% means that its availability is high.
Quality of Criteria for Consumer Health Information | 12 week
  Quality of Criteria for Consumer Health Information scale is to be used in the assessment of the content and quality of educational material. Quality of Criteria for Consumer Health Information consists of 15 key questions plus an overall quality rating. The low total score indicates a poor quality and the high score indicates a good quality. The minimum score to be taken from the scale is 15 and the maximum score is 75.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül İşler Dalgıç, Professor, Study Director — Akdeniz University
Locations (1):
- Süleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Research article
Supporting Information: CSR
Time Frame: 2020-2021
Access Criteria: Open access